CLINICAL TRIAL: NCT07043036
Title: Randomized Controlled Trial Comparing a Strategy Based on Continuous Monitoring at Home Using a Digital Remote Patient Monitoring Solution to Reference Standard in Patients With IBD Initiating an Advanced Therapy or Undergoing a Substantial Change in Their Advanced Therapy.
Brief Title: Randomized Controlled Trial Comparing Remote Patient Monitoring vs Standard Care in IBD Patients Initiating or Changing Advanced Therapy
Acronym: GC-102
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Resilience (Industry)
Collaborators: Sanoia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GC-102; 2024-A02005-42 (ID RCB) (Other: Agence Nationale de Sécurité du Médicament (ANSM))
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: IBD
Keywords: Remote Patient Monitoring; Digital medicine; GutyCare; Resilience; PRO; Patient-reported Outcomes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Treatment (Experimental)
  Interventions: Device: GutyCare
- Control (No Intervention)

INTERVENTIONS:
Device: GutyCare — Device : GutyCare The participants will use GutyCare remote patient monitoring.
  Arms: Intervention/Treatment

SUMMARY:
This clinical trial aims to evaluate whether GutyCare, a digital remote patient monitoring (RPM) solution, can enhance organizational outcomes while maintaining non-inferior clinical results in patients with inflammatory bowel disease (IBD) who are initiating or undergoing significant modifications in advanced therapy.

The study compares standard care to an intervention involving the use of GutyCare, a mobile application that collects patient-reported outcomes related to symptoms.

When clinically significant symptoms are identified, alerts are transmitted to the care team, facilitating timely and personalized therapeutic adjustments.

DETAILED DESCRIPTION:
GutyCare is a digital medical device (dMD, CE marked, class IIa) that enables the remote monitoring of patients diagnosed with Inflammatory Bowel Disease (IBD). GutyCare is a software medical device prescribed by gastroenterologists to collect electronic patient-reported outcomes (ePRO). The workflow of GutyCare includes the following steps:

* Collection of ePRO
* Intelligent analysis and alerts
* Adapted care

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Inflammatory bowel disease, either Crohn's disease or ulcerative colitis, at least 3 months before enrolment
* Initiating an advanced therapy (i.e., biologic therapy or small molecule) OR occurrence of a substantial change in the treatment of the disease.
* Active disease.

Exclusion Criteria:

* Patients with altered intestinal continuity or function due to major abdominal surgery (e.g., stoma, extensive resection, anastomosis), uncontrolled intra-abdominal abscess, or active perianal disease.
* Patients for whom digestive surgery is expected during the study period.
* Patients unable or unwilling to use or already using GutyCare.
* Vulnerable individuals as defined by French law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of on-site IBD-related visits | 12 months

SECONDARY OUTCOMES:
Clinical remission without corticosteroids | 12 months
Patients' disease activity | 12 months
  PRO-2
Improvement in quality of life | 12 months
  SIBDQ

OTHER OUTCOMES:
Experience from patients | 12 months
  Dedicated questionnaire for patients.
Experience from HCP | 12 months
  Dedicated questionnaire for HCP.